CLINICAL TRIAL: NCT02988167
Title: Introducing and Evaluating Extubation AdvisorTM: A Pilot Phase I Observational Study of a Novel Clinical Decision Support Tool to Improve Extubation Decision-making in the Intensive Care Unit
Brief Title: Introducing and Evaluating Extubation Advisor
Acronym: EA
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20160740-01H
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Intubation
Keywords: Spontaneous Breathing Trial (SBT); Extubation Decision Support Tool; Extubation; Extubation Readiness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Knowing when to liberate critically ill patients from mechanical ventilation (i.e. extubation) is of great importance as both prolonged ventilation and failed extubation are associated with increased morbidity, mortality & costs. The study objective is to improve the safety of extubation by harnessing hidden information contained in the patterns of variation of heart and respiratory rate measured over intervals-in-time.

DETAILED DESCRIPTION:
As a standard of care for patients who are intubated in the ICU; to assess ability to be extubated, a Spontaneous Breathing Trial (SBT) is performed, where the level of ventilator support is reduced, and patient's response is observed to predict if they will tolerate extubation.

Spontaneous breathing trials (SBTs) are standard of care in assessing extubation readiness; however, there are no universally accepted guidelines regarding their precise performance and reporting.

Given that health is associated with a high degree of variation of physiologic parameters (e.g. heart and respiratory rate), and illness & stress are associated with a loss of variability, the investigators have demonstrated that maintaining a high level of heart rate (HRV) and respiratory rate variability (RRV) prior to and throughout the Spontaneous Breathing Trial (SBT) will predict successful extubation, and a reduction in heart rate (HRV) and respiratory rate variability (RRV) predicts extubation failure.

Research to date has already demonstrated the added prognostic value and the investigators have derived a predictive model based on continuous monitoring of respiratory rate variability (RRV). The investigators are now poised to evaluate Extubation Advisor (EA) software with the overall goal to transform monitoring and improve care.

This study is a mixed methods, pilot phase I observational study of the clinical implementation of a novel clinical decision support product, Extubation Advisor.TM In this study the investigators will evaluate the feedback of RTs as well as the feedback of MDs post-treatment (extubation) decision.

Questionnaires will be sent to Respiratory Therapists (RT's) and Medical Doctors (MD's) to solicit feedback on the electronic Spontaneous Breathing Trial (SBT) Case Report Form (CRF) and the Extubation Advisor TM (EA) report. All questionnaires will be answered based on a rating scale of 1-5 where 1 is unacceptable and 5 is excellent.

As this proposed study is observational and has no impact on patient care/outcomes, and to avoid bias associated with requiring consent, the investigators believe this study represents one of the limited circumstances under which waived consent may be permitted.

ELIGIBILITY:
Inclusion Criteria:

1. patients who have been or are expected to be on mechanical ventilation for > 48 hours in total prior to extubation,
2. patients who are ready for Spontaneous Breathing Test (SBT) for assessment for extubation,
3. the patients who are able to tolerate pressure support ventilation ≤ 14 cm H2O (SpO2 ≥ 90% with FiO2 ≤ 40% and PEEP 10 ≤ cm H20,
4. patients who are hemodynamically stable (off vasopressors or on low levels of vasopressors: phenylephrine < 50 ug/min; norepinephrine < 5 ug/min; dobutamine < 5 ug/kg/min; milrinone< 0.4 ug/kg/min),
5. patients whose neurological status is stable (no deterioration in the last 24 hrs, intact respiratory drive and ICP <20),
6. patients who have intact airway reflexes (adequate cough with suctioning and a gag reflex), and
7. patient who are in normal sinus rhythm at the time of the SBT (no pacemaker).

Exclusion Criteria:

1. patients who have "do not re-intubate" order documented on their chart or if withdrawal of life support is anticipated,
2. patients who have a tracheostomy,
3. patients who suffer from known or suspected severe myopathy or neuropathy (i.e. myasthenia gravis, Guillain-Barré syndrome) or quadriplegia,
4. patients who have been previously extubated during the same ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being considered for extubation in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Introduce Extubation Advisor TM (EA) | 1 year
  Introduce Extubation Advisor TM (EA) in an observational study in patients being evaluated for extubation, specifically by: (i) engaging RTs to ensure waveform (EKG, CO2) monitoring is in place during spontaneous Breathing Trials (SBTs) and enter clinical data and assessment into the EA data entry screens, (ii) providing RTs and MDs with the EA report at least 48 hours after extubation.
Evaluate Respiratory Therapist (RTs) feedback on the Extubation Advisor TM (EA) | 1 year
  Evaluate: quality and completeness of data elements and process of data entry, integration with existing RT clinical practice and workflow, time to completion of data entry, 48 hours post extubation/treatment decision obtain RT feedback on quality and overall impression of the report.
Evaluate Intensivist (MD) feedback on the Extubation Advisor TM (EA) Report | 1 year
  Evaluate quality and completeness of report, ease of integration into existing MD clinical practice and workflow, overall impression and potential impact on decision making.
Evaluate technical feasibility of future real-time implementation of Extubation Advisor TM (EA) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Sarti, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarti AJ, Zheng K, Herry CL, Sutherland S, Scales NB, Watpool I, Porteous R, Hickey M, Anstee C, Fazekas A, Ramsay T, Burns KE, Seely AJ; Canadian Critical Care Trials Group. Feasibility of implementing Extubation Advisor, a clinical decision support tool to improve extubation decision-making in the ICU: a mixed-methods observational study. BMJ Open. 2021 Aug 12;11(8):e045674. doi: 10.1136/bmjopen-2020-045674. PMID 34385234